CLINICAL TRIAL: NCT02939872
Title: Optimal Duration of Antiplatelet Therapy After Bioresorbable Vascular Scaffold Implantation to Reduce Late Coronary Arterial Thrombotic Events: BVS-LATE Trial
Brief Title: Optimal Duration of Antiplatelet Therapy After Bioresorbable Vascular Scaffold Implantation to Reduce Late Coronary Arterial Thrombotic Events
Acronym: BVS LATE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seung-Jung Park (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, professor, Division of Cardiology, Department of Internal Medicine, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMCCV2016-23
Record Dates: First submitted 2016-10-18; First posted 2016-10-20 (Estimated); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Percutaneous Transluminal Coronary Angioplasty; Coronary Disease
Keywords: DAPT; BVS; Bioresorbable Vascular Scaffold; Dual Antiplatelet Therapy
MeSH Terms: conditions — Coronary Disease | interventions — Aspirin; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DAPT (Experimental): Dual antiplatelet therapy : aspirin and clopidogrel
  Interventions: Drug: aspirin and clopidogrel
- Clopidogrel only (Active Comparator): Clopidogrel monotherapy
  Interventions: Drug: Clopidogrel only

INTERVENTIONS:
Drug: aspirin and clopidogrel — at the discretion of investigator
  Arms: DAPT
Drug: Clopidogrel only — at the discretion of investigator
  Arms: Clopidogrel only

SUMMARY:
The purpose of this study is to evaluate optimal duration of antiplatelet therapy after Bioresorbable Vascular Scaffold implantation to reduce late coronary arterial thrombotic events.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women at least 19 years of age
2. Patients undergoing dual- or triple-antiplatelet therapy at least 12-14 months after PCI with BVS
3. Among the participants underwent PCI with BVS, event-free patients who survived the first 12 months without death, serious MI, stroke, repeat revascularization or major bleeding (except non-significant peri-procedural MI)
4. The patient or guardian agrees to the study protocol and the schedule of clinical follow-up, and provides informed, written consent, as approved by the appropriate Institutional Review Board/Ethical Committee of the respective clinical site.

Exclusion Criteria:

1. Contraindication to antiplatelet therapy
2. If the physician believes that the patient need continuation of dual anti-platelet therapy because of comorbidities (ACS, peripheral vascular disease, significant carotid disease, etc.)
3. Continuous administration of clopidogrel is impossible due to comorbidities of the patient (major bleeding history, bleeding diathesis)
4. Cardiac co-morbid conditions are present with life expectancy <1 year or that may result in protocol non-compliance (per site investigator's medical judgment).
5. Pregnancy test positive (hCG test is performed before randomization in all fertile women)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2017-03-09 (Actual); Primary Completion 2021-05-09 (Actual); Study Completion 2024-06-03 (Actual)

PRIMARY OUTCOMES:
composite event of death, myocardial infarction, or stroke | 1 year

SECONDARY OUTCOMES:
Death | 5 years
  all cause death or cardiac death
Myocardial Infarction | 5 years
Stroke | 5 years
  cerebral ischemic or hemorrhage
Target Vessel Revascularization | 5 years
Target Lesion Revascularization | 5 years
Stent thrombosis | 5 years
Bleeding | 5 years

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Asan Medical Center, Seoul, Songpa-gu
  - Chonnam National University Hospital, Gwangju

IPD SHARING:
Plan to Share IPD: Undecided